CLINICAL TRIAL: NCT02106936
Title: Depotentiation in Focal Hand Dystonia Patients
Brief Title: Depotentiation in People With Focal Hand Dystonia
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: Prachaya Srivanitchapoom, MD (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140070; 14-N-0070
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06-20

CONDITIONS: Focal Dystonia; Healthy Volunteers
Keywords: Focal Hand Dystonia; Depotentiation; Transcranial Magnetic Stimulation (TMS); Rapid Paired Associative Stimulation; Healthy Volunteer
MeSH Terms: conditions — Dystonic Disorders; Dystonia, Focal, Task-Specific

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Background:

- Focal hand dystonia (FHD) causes muscles to contract, leading to abnormal movements or postures. Musicians, writers, and athletes often get it. Researchers want to study how patients with this condition learn, a process of the brain that depends on a property called plasticity.

Objective:

- To study brain plasticity in people with FHD.

Eligibility:

* Right-handed adults 18 years and older with FHD.
* Healthy, right-handed adult volunteers.

Design:

* Participants will be screened with medical history, physical exam, pregnancy test, and questionnaire about their right-handedness.
* Participants will have 2 study visits on 2 different days.
* Participants will sit in a chair and have up to 30 Transcranial Magnetic Stimulation (TMS) pulses on the left side of the head. A brief electrical current passes through a wire coil on the scalp. They will hear a click and may feel a pulling on the skin or muscle twitches. They may have to keep their eyes open and remain alert, tense certain muscles, or perform simple finger movements.
* Forty more pulses, with 10 seconds between, will be given on the left side of the head. Some will be small, some big.
* Researchers will measure muscle response through small electrodes taped to the right hand.
* A cloth cap will be put on the participant s head. Researchers will write on tape on the cap.
* Participants will have the r-PAS. An electrical stimulator will be placed on the nerve at the right wrist. Repeated magnetic pulses will be delivered in trains or short bursts together with electrical stimulation of nerve. Participants will receive up to 840 pulses.
* Participants will be contacted after a few days for a follow-up check.

DETAILED DESCRIPTION:
Objectives:

Primary objectives:

To explore the proper parameters creating a long-term depression (LTD)-like effect and depotentiation (DePo) by using rapid paired associative stimulation (rPAS) in focal hand dystonia (FHD) patients

Sample Size and Population:

We plan to recruit 28 healthy volunteers (HVs) and 28 FHD patients from the Movement Disorders and Botulinum Toxin (BoNT) clinics of HMCS.

Design:

Phase 1 deals with HVs while phase 2 deals with FHD patients. We will complete phase 1 before starting phase 2. Each phase is composed of 2 experiments. In phase 1, experiments 1 and 2 will create the LTD-like effect and DePo in HVs and in phase 2, experiments 3 and 4 will elicit the LTD-like effect and DePo in FHD patients. We will use regression analysis to show that the motor evoked potential (MEP) amplitude declines after eliciting the LTD-like effect and DePo.

Outcome measurements:

Primary outcome:

Determining the parameters for creating the LTD-like effect and DePo in HVs and FHD using rPAS

Secondary outcome:

Measuring the percent change of the MEP amplitude after applying the proper stimulus parameters causing an LTD-like effect and DePo in both HVs and FHD.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must be 18 years or older
* Must be right-handed
* FHD includes only writer s cramp
* Must be able to provide consent
* No open scalp wounds or scalp infections.
* Agrees to not drink caffeine or alcohol for 48 hours before study session.

EXCLUSION CRITERIA:

* Has used illegal drugs within the past 6 months based on history. The intent is to exclude those with drug use that may affect study results. Participants who appear to be intoxicated at the time of testing will be rescheduled.
* Has more than 7 alcoholic drinks a week in the case of a woman and 14 alcoholic drinks a week in the case of a man.
* Abnormal findings on neurologic exam (other than dystonia in patient group)
* Has had a brain tumor, a stroke, head trauma, epilepsy or a history of seizures.
* Has major depression or any major mental disorders (axis I disorders)
* Has a neurologic disorder other than dystonia
* Has had a head injury where there was a loss of consciousness for more than a few seconds.
* Has metal in the body, such as a cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain, cochlear implants, or metal fragments in the eye,
* Has known hearing loss.
* Pregnancy and lactation
* Taking any medication that acts as a central nervous system stimulant or that is known to lower seizure threshold, including, imipramine, amitriptyline, doxepine, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, (MDMA, ecstasy), phencyclidine (PCP, angel s dust), ketamine, gamma-hydroxybutyrate (GHB), alcohol, theophylline, mianserin, fluoxetine, fluvoxamine, paroxetine, sertraline, citalopram, reboxetine, venlafaxine, duloxetine, bupropion, mirtazapine, fluphenazine, pimozide, haloperidol, olanzapine, quetiapine, aripiprazole, ziprasidone, risperidone, chloroquine, mefloquine, imipenem, penicillin, ampicillin, cephalosporins, metronidazole, isoniazid, levofloxacin, cyclosporin, chlorambucil, vincristine, methotrexate, cytosine arabinoside, BCNU, lithium, anticholinergics, antihistamines, and sympathomimetics.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03-05; Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Motor evoked potential amplitude | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Centonze D, Costa C, Rossi S, Prosperetti C, Pisani A, Usiello A, Bernardi G, Mercuri NB, Calabresi P. Chronic cocaine prevents depotentiation at corticostriatal synapses. Biol Psychiatry. 2006 Sep 1;60(5):436-43. doi: 10.1016/j.biopsych.2005.11.018. Epub 2006 Feb 14. PMID 16476411
- [Background] Di Lazzaro V, Pilato F, Dileone M, Profice P, Oliviero A, Mazzone P, Insola A, Ranieri F, Meglio M, Tonali PA, Rothwell JC. The physiological basis of the effects of intermittent theta burst stimulation of the human motor cortex. J Physiol. 2008 Aug 15;586(16):3871-9. doi: 10.1113/jphysiol.2008.152736. Epub 2008 Jun 19. PMID 18566003
- [Background] Figiel GS, Epstein C, McDonald WM, Amazon-Leece J, Figiel L, Saldivia A, Glover S. The use of rapid-rate transcranial magnetic stimulation (rTMS) in refractory depressed patients. J Neuropsychiatry Clin Neurosci. 1998 Winter;10(1):20-5. doi: 10.1176/jnp.10.1.20. PMID 9547462